CLINICAL TRIAL: NCT05349409
Title: A Phase Ⅰb/Ⅱ Clinical Study on the Dosage Exploration and Efficiency Expansion of SHR-A1811 for Injection in Combination With Fluzoparib Capsule in HER2-Expressing Advanced Solid Tumors of Patients
Brief Title: A Trial of the Combination of SHR-A1811 and Fluzoparib in HER2-Expressing Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-Ⅱ-201
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — fluzoparib

STUDY DESIGN:
Intervention Model Description: SHR-A1811 for Injection in combination with Fluzoparib Capsule.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): SHR-A1811, Fluzoparib
  Interventions: Drug: SHR-A1811; Drug: Fluzoparib Capsule

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811 for Injection: Given IV.
Drug: Fluzoparib Capsule — Fluzoparib Capsule: Given PO.
  Other Names: SHR-3162

SUMMARY:
The study is being conducted to evaluate safety, tolerability and preliminary efficacy of SHR-A1811 for Injection in combination with Fluzoparib Capsule for HER2-expressing advanced solid tumors of patients. To explore the reasonable dosage of dosage regimen of combination therapy for HER2-expressing advanced malignant tumors of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years at the time of signing the ICF.
2. At least one measurable lesion that meets RECIST 1.1 criteria in case of solid tumors.
3. An Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1.
4. Life expectancy ≥12 weeks.
5. Adequate organ functions as defined.
6. Swallow the drug pills normally.

Exclusion Criteria:

1. patients with active meningeal metastasis, or brain metastasis without surgical treatment or radiotherapy.
2. Cancerous ascites and pleural effusion with clinical symptoms, which need puncture and drainage.
3. Prior malignancy (other than current malignant tumor) within 5 years before the first dose of study treatment.
4. History of autoimmune diseases.
5. Not well controllable and serve cardiovascular disease.
6. Prior lung disease with clinical significance.
7. Occurrence of ≥ grade 2 of bleeding event within 4 weeks before the first dose, or currently receiving the anticoagulation.
8. Active Hepatitis B and Hepatitis C; or serve infection with medication control.
9. The grade of toxicity from the prior anti-cancer therapy not decrease to ≤ 1.
10. Occurrence of intestinal obstruction and gastrointestinal perforation within 3 months before the first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity | first dose of study medication up to 21 days
  Dose Limited Toxicity of SHR-A1811 for Injection in combination with Fluzoparib Capsule in Dose Exploration Period
Recommended phase II dose | first dose of study medication up to 21 days
  The Recommended phase II dose of SHR-A1811 for Injection in combination with Fluzoparib Capsule in Dose Exploration Period
ORR | from the date of the first dose to the date of disease progression evaluated based on RECIST v1.1 criteria, or initiation of other anti-tumor treatment, whichever occurs first, up to 6 months
  Objective Response Rate, Efficacy endpoints of SHR-A1811 for Injection in combination with Fluzoparib Capsule in HER2-Expressing Advanced Solid Tumors of Patients in indication expansion period

SECONDARY OUTCOMES:
DoR | from the date of the firstly documented tumor response (evaluated based on RECIST v1.1 criteria) to the date of the firstly documented disease progression (evaluated based on RECIST v1.1 criteria) or the date of death for any reason, up to 6 months
  Duration of response, Efficacy endpoints of SHR-A1811 for Injection in combination with Fluzoparib Capsule in HER2-Expressing Advanced Solid Tumors of Patients
DCR | from the date of the first dose to the date of the firstly documented disease progression (evaluated based on RECIST v1.1 criteria) or the date of death for any reason, up to 6 months
  Disease control rate, Efficacy endpoints of SHR-A1811 for Injection in combination with Fluzoparib Capsule in HER2-Expressing Advanced Solid Tumors of Patients
TTR | from the date of the first dose to the date of treatment termination, up to 6 months
  Time to Recovery, Efficacy endpoints of SHR-A1811 for Injection in combination with Fluzoparib Capsule in HER2-Expressing Advanced Solid Tumors of Patients
PFS | from the date of the first dose to the date of the firstly documented disease progression (evaluated based on RECIST v1.1 criteria) or the date of death for any reason, up to 6 months
  Progression-free survival, Efficacy endpoints of SHR-A1811 for Injection in combination with Fluzoparib Capsule in HER2-Expressing Advanced Solid Tumors of Patients
OS | from the date of the first dose to the date of death for any reason, up to 100 months
  Overall survival, Efficacy endpoints of SHR-A1811 for Injection in combination with Fluzoparib Capsule in HER2-Expressing Advanced Solid Tumors of Patients
12 months' survival rate | from the date of the first dose up to 12 months
  Efficacy endpoints of SHR-A1811 for Injection in combination with Fluzoparib Capsule in HER2-Expressing Advanced Solid Tumors of Patients
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) | from signature completion of ICF to 30 days after the last dose or to the beginning of the new anti-cancer therapy, up to 6 months
  Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
The occurrence rate of dose titration due to AE related with study medication | from signature completion of ICF to 30 days after the last dose or to the beginning of the new anti-cancer therapy, up to 6 months
  The occurrence rate of dose interruption, dose decrease and dose termination because of study drug related toxicity during the study
Cmin | 10 min before first dose of Fluzoparib Capsule in C1D8 to 10 min before first dose of Fluzoparib Capsule in C8D1
  PK concentration of Fluzoparib Capsule
C3h | 3 hour after first dose of Fluzoparib Capsule in C2D1
  PK concentration of Fluzoparib Capsule
AUC0-t | the date of first dose to 30 days after last dose
  PK parameters of SHR-A1811 for Injection
Cmin | the date of first dose to 30 days after last dose
  PK parameters of SHR-A1811 for Injection
Cmax | the date of first dose to 30 days after last dose
  PK parameters of SHR-A1811 for Injection
ADA | the date of first dose up to 90 days after last dose
  Anti-drug antibody, Immunogenicity of SHR-A1811 for Injection
NAb | the date of first dose up to 90 days after last dose
  Neutralizing Antibody, Immunogenicity of SHR-A1811 for Injection

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided